CLINICAL TRIAL: NCT06945315
Title: Robotic-Assisted Laparoscopic Prostatectomy (RALP) and SAFE (Saline Assisted Fascial Engorgement) Nerve Preservation Guided by Micro-ultrasound: A Phase III RCT
Brief Title: SAFE Nerve Sparing Guided by Micro-ultrasound (MUS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ashutosh Kumar Tewari, Professor and System Chair, Milton and Carroll Petrie Department of Urology. Director of Center of Excellence for Prostate Cancer at the Tisch Cancer Institute, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY-22-01522
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: Robotic-Assisted Laparoscopic Prostatectomy (RALP); SAFE (Saline assisted fascial engorgement)
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors (physician associate/physician assistant or Nurse practitioner) will be blinded from the study arm allocated. While investigators cannot be blinded due to the nature of the intervention, implementation of allocation concealment will minimize the chance of potential allocation biases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RALP with SAFE Technique (Experimental): Erectile function recovery will be evaluated for patients receiving Robotic-Assisted Laparoscopic Prostatectomy (RALP) + SAFE (Saline assisted fascial engorgement).
  Interventions: Procedure: RALP (Robotic-assisted radical prostatectomy); Drug: SAFE (Saline assisted fascial engorgement)
- RALP without SAFE Technique (Active Comparator): Erectile function recovery will be evaluated for patients receiving Robotic-Assisted Laparoscopic Prostatectomy (RALP) without SAFE (Saline assisted fascial engorgement).
  Interventions: Procedure: RALP (Robotic-assisted radical prostatectomy)

INTERVENTIONS:
Procedure: RALP (Robotic-assisted radical prostatectomy) — Robotic-assisted radical prostatectomy (RALP) is a standard surgical procedure for managing localized prostate cancer that focuses on prostate anatomy and surrounding structures to enable personalized surgeries. The procedure incorporates nerve-sparing techniques through careful dissection of the neurovascular bundle and can use a thermal and traction-free dissection to improve functional outcomes, particularly erectile function.
Drug: SAFE (Saline assisted fascial engorgement) — SAFE (Saline assisted fascial engorgement) an innovative technique to achieve enhanced nerve-sparing outcomes among patients undergoing robot-assisted laparoscopic radical prostatectomy (RALP). Essentially a new method of hydro dissection, SAFE involves an injection of 30 cc of normal saline solution between the layers of the periprostatic fascia after early release of the neurovascular bundle. This injection effectively pushes the nerves away from the prostate, enabling a dissection of the prostate that is atraumatic vis a vis the neural hammock.
  Arms: RALP with SAFE Technique

SUMMARY:
Robotic-assisted radical prostatectomy (RALP) has become the standard of care in the management of localized prostate cancer. However, post-prostatectomy erectile dysfunction (ED) and urinary incontinence still pose a challenge that adversely affects the patient's quality of life. Hydrodissection (HD) was introduced in 1987 in the medical field and it was tested for the first time during a retropubic radical prostatectomy back in 2005. Since then, research has indicated an improvement in erectile function results, presumably because of a less traumatic neural dissection and a decreased risk of neuropraxia. In an effort to achieve a balance between oncological excision and functional preservation, prostate surgery is evolving to incorporate intraoperative real-time evaluation of extracapsular extension. Recently, a micro-ultrasound operating at 29 MHz has been introduced. It provides a resolution down to 70 μ to assess the glandular pattern and cellular density of the prostatic tissue. Given the experience in more than a thousand cases with this technology, and the growing literature showing promising results in the detection and staging of prostate cancer; the researchers decided to implement this tool as guidance for hydrodissection of the layers of the lateral prostatic fascia.

Robotic-Assisted Laparoscopic Prostatectomy and SAFE (Saline assisted fascial engorgement) nerve preservation guided by Microultrasound (MUS) is a prospective randomized controlled trial designed to evaluate the impact of normal saline solution hydrodissection (HD) on erectile function outcomes after RALP. This innovative approach consists of a transrectal ultrasound-guided HD using a high-resolution Microultrasound (MUS) (ExactVu micro-ultrasound, Exact Imaging, Markham, Canada). The technique will be applied to those patients who undergo grade 1, 2, or 3 NS approach taking into account the grading system proposed by Tewari et al.

The hypothesis is that the SAFE technique could minimize the risk of a traumatic neurovascular bundle dissection while assessing the prostatic capsule integrity with a high-resolution MUS. The researchers also hypothesize that the use of SAFE along with RALP will optimize the post-surgery recovery of erectile function.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at the time of consent.
* Men who are potent (SHIM ≥ 17) and sexually active, who are planned to undergo a grade 1, 2, or 3 nerve-sparing approaches, as per the grading system during RALP.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects who are candidates for salvage RALP
* Subjects on androgen deprivation therapy (ADT)
* Subjects in whom PDE5 inhibitors are contraindicated

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since this is a prostate cancer study, only male candidates are eligible for the study.
Enrollment: 196 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2027-07-14 (Estimated); Study Completion 2027-07-14 (Estimated)

PRIMARY OUTCOMES:
Sexual Health Inventory for Men (SHIM) | Baseline (Week 0), 6 weeks, 3-months, 6-months, 12-months and 24-months following surgery
  The Sexual Health Inventory for Men (SHIM) is a five-question, abbreviated, validated questionnaire derived from the International Index of Erectile Function questionnaire. It is widely used by urologists to evaluate efficacy of ED treatments. It is graded on a scale of 1-25, with higher scores indicating no signs of erectile dysfunction.

SECONDARY OUTCOMES:
The Erection Hardness Score (EHS) | Baseline (Week 0), 6 weeks, 3-months, 6-months, 12-months and 24-months following surgery
  The Erection Hardness Score (EHS) is tool used to evaluate and monitor the severity of ED. It is a four-point scale (1-4), with a score of 4 indicating a completely hard and fully rigid erection. Higher score indicates better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Kumar Tewari, MBBS, MCh, FRCS (Hon.), Principal Investigator — Study Principal Investigator
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in ISMMS data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (to be determined).